CLINICAL TRIAL: NCT01433068
Title: An Open-Label, Single Arm, Feasibility And Safety Phase I Study With NBTXR3 Intratumor Implantation (By Injection) And Activated By External Beam Radiation Therapy In Patients With Soft Tissue Sarcoma Of The Extremity And Trunk Wall
Brief Title: NBTXR3 Crystalline Nanoparticles and Radiation Therapy in Treating Patients With Soft Tissue Sarcoma of the Extremity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanobiotix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBTXR3-101; ID RCB : 2011-A00342-39 (Other: Afssaps)
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Adult Soft Tissue Sarcoma
Keywords: Adult Soft Tissue Sarcoma of the extremities and Trunk wall
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NBTXR3 (Experimental)
  Interventions: Device: NBTXR3

INTERVENTIONS:
Device: NBTXR3 — One intratumor implantation by injection

SUMMARY:
RATIONALE: Radiation therapy given before surgery of soft tissue sarcoma decreases the size of the tumor mass and the presence of malignant cells in its peripheral region. NBTXR3 and radiation therapy may kill more cancer cells and increase the tumor shrinkage rendering surgery more feasible or easier and achieve better local control of the tumor.

PURPOSE: This Phase I trial aims at evaluating the feasibility of the NBTXR3 injection in the tumor, safety and the adequate dose of NBTXR3 when given with radiation therapy.

DETAILED DESCRIPTION:
Patients will receive a single intratumor injection of NBTXR3 on day 1 and will receive external beam radiotherapy starting on day 2 up to completion of 5 weeks, 5 days a week of treatment (50Gy, 2Gy/fraction). Then, all patients will undergo surgical resection of the tumor 5 weeks later and will be followed for wound healing and toxicity assessment. A visit of end of treatment will take place approximately 3-4 weeks after surgery. Patients will be followed for evaluation of their disease status and adverse events every 8 weeks until the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older
* Soft tissue sarcoma of the extremity or trunk wall, or localized in the posterior region of the neck (i.e., coronal section passing through the posterior limit of the ear)
* Locally advanced soft tissue sarcoma,candidate to radiotherapy

  * Primary tumor or,
  * Relapsed tumor, localized out of already irradiated area or,
  * Sarcomas secondary to previous irradiation exposure due to other primary cancer
* WHO performance score 0 to 2
* Adequate function of Bone marrow:
* Adequate renal function
* Adequate liver function
* All female patients of childbearing potential must have a negative serum/urinary pregnancy test

Exclusion Criteria:

* Written Informed Consent not obtained, signed and dated
* Patients with the following histological type: Gastrointestinal Stromal Tumors (GIST), embryonal or alveolar rhabdomyosarcoma, Ewing's sarcoma, osteosarcoma or chondrosarcoma, Kaposi's sarcoma, primitive neuroectodermal tumor or dermatofibrosarcoma protuberans
* Soft tissue sarcoma of the trunk wall localized in the abdominal region, i.e. the region defined cranially by the xiphoid process of the sternum and the costal margins, and caudally by the line joining the anterior superior iliac spines, both limited by the perpendicular lines crossing both nipples
* Angiosarcoma of the trunk wall because of its diffuse frontier
* Metastatic disease (CT-scan verification) with survival expectation < 6 months
* Concurrent treatment with any other anticancer therapy
* Absence of histologically or cytologically proven cancer at the first diagnosis
* Previous neoadjuvant chemotherapy treatment given as an upfront of the current treatment line
* Previous radiation therapy in relapse site of the soft tissue sarcoma (no radiation re-challenge is permitted)
* Moderate and severe liver dysfunction
* Hemolytic anemia
* Autoimmune disease
* Complete initial work up earlier than 4 weeks prior to patient registration
* Patients unable to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Patients participating in another clinical investigation at the time of signature of the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the feasibility of the intratumor injection of NBTXR3 | 6 months
  - To evaluate the feasibility of NBTXR3 given as intratumor implantation (by injection) and activated by external beam radiation in patients with soft tissue sarcoma of the extremity and trunk wall
Assessment of the safety profile and determination of early dose limiting toxicity | 20 months
  - To assess the safety profile and determine the early dose limiting toxicity (DLT) of NBTXR3 intratumor implantation (by injection) and activated by external beam radiation

SECONDARY OUTCOMES:
Evaluation of the anti-tumor activity of NBTXR3 in terms of pathological Response (pR) | 20 months
  - To evaluate the anti-tumor activity of NBTXR3 implanted within the tumor (by injection) at Day 1 and activated 24 hours later by external beam radiation therapy in terms of pathological Response (pR)
Evaluation of the Response Rate (RR) of NBTXR3 as per RECIST | 20 months
  - To evaluate the Response Rate (RR) of NBTXR3 implanted within the tumor (by injection) at Day 1 and activated 24 hours later by external beam radiation therapy as per RECIST
Characterization of the body kinetic profile of NBTXR3 | 20 months
  - To characterize the body kinetic profile of NBTXR3 implanted within the tumor (by injection) at Day 1 and Day 2 before its activation by radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie BONVALOT, MD-PhD, Principal Investigator — Head of Surgery Division; Guy KANTOR, MD-PhD, Principal Investigator — Head of Radiotherapy Department
Locations (2):
- France (2):
  - Institut Bergonie, Bordeaux
  - Institut Gustave Roussy, Villejuif